CLINICAL TRIAL: NCT04256759
Title: Dupilumab for the Treatment of Moderate to Severe Chronic Hepatic Pruritus: an Open-Label, Single-Arm, Exploratory Study
Brief Title: Dupilumab for the Treatment of Moderate to Severe Chronic Hepatic Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jason Sluzevich MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-002757
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pruritus
Keywords: Dupilumab
MeSH Terms: conditions — Pruritus | interventions — dupilumab; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dupilumab (Experimental): Subcutaneous (SC) dupilumab selected for this study is 300 mg every 2 weeks for 18 weeks.
  Interventions: Drug: Dupilumab 300Mg Solution for Injection

INTERVENTIONS:
Drug: Dupilumab 300Mg Solution for Injection — Subcutaneous (SC) dupilumab selected for this study is 300 mg every 2 weeks for 18 weeks.
  Other Names: Dupixent

SUMMARY:
To investigate the potential efficacy of dupilumab in the treatment of moderate to severe chronic hepatic pruritus.

DETAILED DESCRIPTION:
This is a 22-week (2 week screening, 18-week treatment period followed by a 2 week followup), phase II, open label, exploratory study to investigate the potential efficacy of FDA approved dupilumab in the treatment of adults with moderate to severe chronic hepatic pruritus. Subjects will be screened at outpatient clinic visit appointments and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained, baseline values will be established and subjects will begin treatment and follow-up for the next 20 weeks. A final visit will be needed for evaluation and questionnaire completion.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects 18 years or older with chronic pruritus of moderate to severe severity in the setting of intrahepatic or extrahepatic cholestatic liver disease. Chronic is defined as greater than 6 weeks of symptom duration. Pruritus severity is based on the peak pruritus numerical rating score of ≥ 4 (moderate severity).
* Documentation of a personally signed and dated informed consent indicating that the subject or their legally acceptable representative has been informed of all pertinent aspects of the trial.
* Willingness and ability to comply with scheduled clinic visits, physical exams, laboratory tests, questionnaires, effective contraception use, and other trial procedures.

Exclusion Criteria:

* Male and/or female subjects under 18 years of age.
* Pruritus due to a primary inflammatory skin dermatosis or other forms of psychogenic pruritus utilizing skin biopsies as needed.
* Pregnant females
* History of intrahepatic cholestasis of pregnancy
* Any form of chronic hepatic pruritus associated with underlying malignancy
* Liver transplant recipients
* Allergy to dupilumab or its ingredients
* Inability to provide informed consent
* Concomitant use of selective opioid antagonists
* Subjects with severe asthma (requiring high-dose inhaled or systemic corticosteroids) will be excluded from the study.
* Patients with known helminth infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sluzevich, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Dupilumab: Subcutaneous (SC) dupilumab selected for this study was 300 mg every 2 weeks for 18 weeks.
  Dupilumab 300Mg Solution for Injection: Subcutaneous (SC) dupilumab selected for this study was 300 mg every 2 weeks for 18 weeks.
Period: Overall Study
Arm/Group | Dupilumab
Started | 9
Completed | 7
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dupilumab
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Pruritus Numerical Rating Score (PRNS)
Description: Pruritus severity is measured using the peak PNRS assessed as a single, self-completed item that assesses the intensity of peak (worst) pruritus during the past 24 hours using the query: "On a scale of 0 to 10, with 0 being 'no itch 'and 10 being 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Measured before and after treatment. Scores range from 0 to 10 with higher scores indicating a worse outcome.
Time Frame: Baseline; 20 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 9
score on a scale | -3.1 (3.9)

2. Secondary Outcome: Change in Weekly Average Peak Pruritus Numerical Rating Score (PRNS) ≥3 From Baseline
Description: Pruritus severity is measured using the peak PNRS assessed as a single, self-completed item that assesses the intensity of peak (worst) pruritus during the past 24 hours using the query: "On a scale of 0 to 10, with 0 being 'no itch 'and 10 being 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Scores range from 0 to 10 with higher scores indicating a worse outcome.
Time Frame: Baseline; week 6,12,18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 9
score on a scale
  Week 6 | -3.2 (3.6)
  Week 12 | -3.5 (3.9)
  Week 18 | -4.1 (4.4)

3. Secondary Outcome: Verbal Rating Scale (VRS) Score
Description: The number of subjects who rated their intensity of pruritus as 0=none, 1=mild, 2-moderate, 3=severe. The verbal rating scale measures the intensity of pruritus. Subjects are asked to rate their pruritus intensity as 0=none; 1= mild; 2=moderate; and 3=severe/intense. Scores range from 0 to 3, with higher scores indicating a worse outcome.
Time Frame: Baseline; week 12,18
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 9
Participants
  Baseline-None | 0
  Baseline-Mild | 0
  Baseline-Moderate | 4
  Baseline-Severe | 5
  Week 12-None | 1
  Week 12-Mild | 4
  Week 12-Moderate | 3
  Week 12-Severe | 0
  Week 18-None | 2
  Week 18-Mild | 4
  Week 18-Moderate | 2
  Week 18-Severe | 0
Statistical Analysis 1: Comparison: Dupilumab; Week 12; Test type: Superiority; p = 0.018, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dupilumab; Week 18; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Chronic Liver Disease Questionnaire (CLDQ) Score
Description: This is a validated 29 question quality life instrument for patients with chronic liver disease evaluating systemic symptoms, fatigue, physical activity, emotional function, and worry. Subjects are asked to respond to each question using the following scale: 6=all of the time; 5=most of the time; 4=a good bit of the time; 3=some of the time; 2=a little of the time; 1=hardly any of the time; and 0=none of the time. Total scores range from 0 to 174 with lower scores indicating better health-related quality of life.
Time Frame: Baseline; 18 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 9
score on a scale | 25.7 (38.7)
Statistical Analysis 1: Comparison: Dupilumab; Test type: Superiority; p = 0.13, t-test, 2 sided

5. Secondary Outcome: Change in 5D Pruritus Score
Description: This is a multidimensional questionnaire designed to assess the degree, duration, direction, disability and distribution of pruritus longitudinally with scoring ranging from 5=no pruritus/well-controlled to 25=severe pruritus/poorly controlled, with higher scores indicating a worse outcome.
Time Frame: Baseline; 18 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 9
score on a scale | -7.3 (4.6)
Statistical Analysis 1: Comparison: Dupilumab; Test type: Superiority; p = 0.006, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 22 weeks.
Description: The adverse event definition used in this study was: An untoward or undesirable experience associated with the use of a medical product (i.e. drug, device, biologic) in a patient or research subject. Adverse events were collected through specific questioning and physical examinations.
Arm/Group | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04256759/Prot_SAP_000.pdf